CLINICAL TRIAL: NCT00399945
Title: A Phase 1, Single-Dose, Open-Label, Two-Way Crossover, Pharmacoscintigraphy Study of Aerosol Delivery Characteristics (Measured by In Vivo Lung Deposition, Nebulization Time, Serum Tobramycin Concentrations, and Pharmacokinetic Parameters) and Safety of Tobramycin Administered for Inhalation by PARI eFlow® Rapid Electronic Nebulizer (No Compressor) vs. PARI LC PLUS (TM) Jet Nebulizer (With Compressor) in Healthy Subjects and in Subjects With Cystic Fibrosis
Brief Title: Tobramycin Inhalation Solution Administered by eFlow Rapid Nebulizer: Scintigraphy Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTBM100B2202
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis, tobramycin, PARI eFlow, PARI LC Plus, nebulizer, pharmacoscintigraphy
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tobramycin

INTERVENTIONS:
Drug: Tobramycin

SUMMARY:
This study assesses the aerosol delivery characteristics (measured by in vivo lung deposition, nebulization time, serum tobramycin concentrations, and pharmacokinetic parameters) and safety of tobramycin inhalation solution administered for inhalation by PARI eFlow rapid electronic nebulizer (no compressor) vs. PARI LC PLUS Jet Nebulizer (with compressor) in healthy subjects and in subjects with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Provide written informed consent prior to the performance of any study-related procedures.
* Be 18 to 65 years of age at screening.
* Weigh within ± 25% of the ideal using the body mass index method.
* Able to comply with all protocol requirements.

Healthy Subjects:

* Be healthy males or non-pregnant, non-breast-feeding healthy females.
* Have an forced expiratory volume in one second (FEV1) of at least 80% of predicted or greater based on age, sex, height, and race based on European Community for Steel and Coal (ECSC) equations

Subjects with Cystic Fibrosis:

* Be chronically colonized with Pseudomonas aeruginosa .
* Have a diagnosis of CF by documented sweat chloride of 60 mEq/L or greater by quantitative pilocarpine iontophoresis test (QPIT) and/or genotype with two identifiable mutations consistent with CF, accompanied by one or more clinical features consistent with CF.
* Have an FEV1 of 25% or more of the predicted value, calculated using ECSC equations based on age, sex, height, and race.
* Able to tolerate a 1-week washout interval with no inhaled tobramycin or other aminoglycoside treatment.
* Be clinically stable in the opinion of the referring investigator at the CF unit.

Exclusion Criteria:

All subjects:

* Participation in a clinical research study within the previous 1 month.
* History of alcohol or drug abuse.
* Positive result for drugs of abuse.
* Regular alcohol consumption in males and females of more than 21 units and 14 units per week, respectively
* Known hypersensitivity to salbutamol.
* Current smoker or smoked within the last 12 months.
* Breath carbon monoxide reading of greater than 10 ppm either at the prestudy medical examination or on a study day prior to dosing.
* Females of childbearing potential, who are pregnant who plan to become pregnant during the course of the study, who are breast feeding, or who are sexually active and either not using a reliable form of contraception or not surgically sterile.
* Clinically significant abnormal biochemistry, hematology, or urinalysis.
* Positive hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV) results.
* Treatment with any investigational drug within 1 month before screening.
* Treatment with loop diuretics within 7 days before study drug administration.
* Serum creatinine or blood urea above the upper limit of normal for sex and age, or an abnormal urine analysis defined as 2+ or greater proteinuria.
* Known local or systemic hypersensitivity to aminoglycosides.

Healthy Subjects:

* Screening FEV1 less than 80% of the predicted value for sex, age, height, and race using ECSC equations
* History of chronic respiratory disorders, including asthma.
* Treatment with tobramycin or other aminoglycosides within 1 week prior to the study.
* History of adverse reaction or allergy to tobramycin or other aminoglycosides.
* History of infantile bronchiolitis or a history or the presence of asthma or wheezy respiration.
* Upper respiratory tract infection (excluding otitis media) within 14 days of the first study day or lower respiratory tract infection within the last 3 months.
* Treatment with any medication that may affect the respiratory tract within 1 week of the first study day and throughout the study (oral contraceptives, Hormone Replacement Therapy [HRT], and paracetamol are permitted);
* Failure to satisfy the Principal Investigator regarding fitness to participate for any other reason.
* Donation of blood within the previous 3 months.
* Treatment with diuretics or history of renal failure.
* Radiation exposure from clinical trials. No subject whose occupational exposure is monitored is eligible to participate in the study.

Subjects with Cystic Fibrosis:

* Screening FEV1 less than 25% of the predicted value for sex, age, height, and race using ECSC equations
* Treatment with inhaled or intravenous aminoglycosides within 7 days before study drug administration.
* Current treatment with inhaled tobramycin delivered by the PARI LC PLUS jet nebulizer who do not have a washout period of at least 1 week before entering the study.
* Hemoptysis more than 60 mL at any time within 30 days before study drug administration.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2006-05

PRIMARY OUTCOMES:
Lung deposition of tobramycin when inhaled using either PARI LC PLUS jet nebulizer or PARI eFlow rapid Electronic Nebulizer

SECONDARY OUTCOMES:
Nebulisation time for inhaling tobramycin using PARI LC PLUS jet nebulizer or PARI eFlow rapid Electronic Nebulizer
Correlation between tobramycin deposition and serum tobramycin concentrations and pharmacokinetics
Safety of tobramycin when inhaled using either PARI LC PLUS jet nebulizer or PARI eFlow rapid Electronic Nebulizer

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Stoke-on-Trent, United Kingdom